CLINICAL TRIAL: NCT03765034
Title: Constraint-Induced Movement Therapy and Occupational Therapy for Perinatal Brachial Plexus Injury: A Randomized Crossover Trial
Brief Title: Constraint-induced Movement Therapy for Perinatal Brachial Plexus Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, julie werner, Clinical Scientist, Children's Hospital Los Angeles
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CCI-10-00255
Record Dates: First submitted 2018-12-03; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Neonatal Brachial Plexus Palsy
MeSH Terms: conditions — Neonatal Brachial Plexus Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Constraint-induced Movement Therapy (Experimental): A passive constraint cast is applied to the participant's unaffected arm to prevent use for 8 weeks.
  Interventions: Behavioral: Constrain-induced Movement Therapy; Behavioral: Usual Occupational Therapy
- Usual Occupational Therapy (Active Comparator): Usual and standard care occupational therapy is administered for 8 weeks.
  Interventions: Behavioral: Usual Occupational Therapy

INTERVENTIONS:
Behavioral: Constrain-induced Movement Therapy — 8-week therapy program utilizing constraint of the unaffected arm
  Arms: Constraint-induced Movement Therapy
Behavioral: Usual Occupational Therapy — 8-week therapy program without constraint of the unaffected arm

SUMMARY:
This study evaluates the addition of constraint-induced movement therapy (CIMT) to usual care occupational therapy in children with perinatal brachial plexus injury. Participants are randomized to receive either the intervention (CIMT) or control first, then cross over to receive the other one.

DETAILED DESCRIPTION:
Children with perinatal brachial plexus injury routinely receive occupational therapy intervention to improve strength and function in their weak or paralyzed arm.

Constraint-induced movement therapy (CIMT) is known to increase upper extremity function in children with weakness or disuse as a result of cerebral palsy. However, it is unknown if this therapy is effective for treating arm weakness or disuse as a result of perinatal brachial plexus injury. The addition of CIMT to usual and standard occupational therapy care is evaluated in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Participant has perinatal brachial plexus injury
* Participant walking at time of study inception
* Ability to cooperate with interventions and assessment
* Participant currently receiving occupational therapy 1+ hour per week and planning to continue for duration of study

Exclusion Criteria:

* Co-morbid diagnosis not related to perinatal brachial plexus injury
* Flaccidity of the involved upper extremity or no observable hand function
* Planned surgery or drug intervention during the study period
* Allergy or intolerance to constraint intervention materials

Ages: 12 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Assisting Hand Assessment 5.0 | change from baseline at 8 weeks and 16 weeks
  Criterion-referenced observational scale of affected hand use during bimanual performance. Each item is score 1-4 (1 = does not do; 2 = ineffective; 3 = somewhat effective; 4 = effective), yielding a Rasch-modeled standardized score between 0 and 100.